CLINICAL TRIAL: NCT02956408
Title: Efficacy of Vitamin D Supplementation in Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Aviva B. Sopher, Assistant Professor of Pediatrics, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAQ9255
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Obesity, Pediatric; Obesity, Childhood; Obesity, Morbid; Vitamin D Deficiency
Keywords: Obesity; Pediatrics; Vitamin D deficiency
MeSH Terms: conditions — Pediatric Obesity; Obesity, Morbid; Vitamin D Deficiency; Obesity | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): Patients in this arm will be prescribed Vitamin D3 2000 IU once a day
  Interventions: Dietary Supplement: Vitamin D3
- High Dose (Experimental): Patients in this arm will be prescribed Vitamin D3 6000 IU once a day
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Patients will be prescribed either 2000 IU or 6000 IU of vitamin D3 per day. They will go to a pharmacy and purchase a vitamin D3 supplement in their preferred form (eg gummy, liquid, chew, tablet, capsule)
  Other Names: Cholecalciferol

SUMMARY:
Vitamin D deficiency is common in the general population in the United States, but is more common in overweight and obese children. Additionally, vitamin D levels are inversely correlated with body mass index, hypertension, inflammatory markers and insulin resistance. There are currently no clear guidelines regarding vitamin D replacement in obese but otherwise healthy children. The Endocrine Society recommends that children with vitamin D deficiency should take 2000 IU once a day for at least 6 weeks; however, they state that obese children may need 2-3 times this dose in order to reach sufficient levels.

The goals of this study are:

1. To determine the prevalence of vitamin D sufficiency (>30 ng/mL), insufficiency (21-29 ng/mL); deficiency (10-19 ng/mL) and severe vitamin D deficiency (<10 ng/dL) in an obese pediatric population (2-11 years) as measured by 25-hydroxyvitamin D.
2. To determine if vitamin D level correlates with percentage body fat by bioelectrical impedance analysis and/or visceral fat by waist circumference in children ages 5 - 11 years.
3. To observe the effect of vitamin D replacement in obese children with vitamin D deficiency using two different replacement dosage levels recommended by the Endocrine Society over three months: 2000 IU once a day (general pediatric dose) vs 6000 IU once a day (suggested obesity dose) in children between the ages of 5 - 11 years.
4. To measure vitamin D levels, bone markers, inflammatory markers and vitamin D binding protein before and after vitamin D supplementation in children between the ages of 5 - 11 years. Analysis will be stratified by degree of obesity (Class I, Class II, Class III) and season.

DETAILED DESCRIPTION:
Study subjects will be obese children between the ages of 2 and 11 years who are being seen at the FIT (Families Improving Health Together) program. As part of their routine care, all patients seen at the FIT program will have weight measured to the nearest 0.1 kilogram by digital floor scale, stature by wall-mounted stadiometer and waist circumference measurements to the nearest 0.1 centimeter. BMI will be calculated as weight in kilograms, divided by height in meters squared (kg/m2). Waist circumference will be measured with a tape measure at the uppermost lateral border of the hip crest (ilium). Percentage body fat will be approximated by bioelectrical impedance analysis. All patients will have 25-hydroxyvitamin D measured, which will be sent to Esoterix Labs (Calabasas Hills, CA) and run by high-pressure liquid chromatography/tandem mass spectrometry (HPLC/MS-MS). Other baseline labs that will be drawn include glucose, insulin, hemoglobin A1c, lipid panel, hepatic function panel and basic metabolic panel. Blood from the initial visit will be banked for future research laboratory testing as part of the overall goal of the FIT program. The research labs that will be run include vitamin D binding protein, osteocalcin, c-telopeptide, P1NP, PTH, IL-6 and TNF-alpha.

Vitamin D prevalence information and baseline labs and anthropometrics will be obtained from all patients who agree to participate in the study; however, bioelectrical impedance analysis will not be performed in patients under 5 years. Patients between the ages of 5 and 11 years who have a 25-hydroxyvitamin D below 21 ng/mL will be invited to participate in vitamin D supplementation portion of the study. These patients will be treated with vitamin D3 supplementation of either 2000 IU once a day or 6000 IU once a day. Dose will be determined by a set dosing schedule. Each provider will be assigned a dosing schedule and dosing schedules that will change every 3 months over 2 years. The dosing schedule can be found in the study documents section. This study design is intended to minimize bias based on provider or season. Eligible patients who agree to participate in the study will purchase the prescribed dose of vitamin D3, which is an over the counter medication. Vitamin D3 is supplied over the counter as drops, liquid, chewable tablets, gummies, tablets or capsules and parents will select the form that is easiest for their child to take. They will supply us with a picture of the vitamin D3 label so that we can ensure they are taking the appropriate dose and form of vitamin D. They will take the prescribed dose every day for three months. Patients will get weekly reminder calls to ensure that they are taking the supplement as prescribed. At the end of three months they will return for their scheduled clinic appointment. Weight, height, waist circumference and percentage body fat will be measured and labs will be redrawn including 25-hydroxyvitamin D glucose, insulin, hemoglobin A1c, lipid panel, hepatic function panel and basic metabolic panel and the research labs described above will be drawn as well. At the end of 3 months if vitamin D is 21 ng/mL or above they will be advised to take vitamin D 1000 IU once a day; if their vitamin D continues to be below 21 ng/mL they will be advised to continue their current dose of vitamin D.

We expect to see on average about 8 new patients per week and we expect that at least 50% of them will have vitamin D level below 21 ng/mL and will be between the ages of 5 and 11 years. Over two years that amounts to 416 prospective study subjects. Dosages selected are based on the Endocrine Society Clinical Practice Guidelines (2011), which state that children with vitamin D deficiency should be treated with 2000 IU of vitamin D once a day; however obese children should be treated with 2-3 times that amount. In total we expect to enroll 192 subjects over two years to the intervention portion of this trial (5 - 11 years) and we expect to enroll a total of 400 subjects to the observational portion (prevalence and associations with lab testing).

Exclusion criteria include the following: Underlying disorder of bone metabolism, chronic renal failure, chronic steroid treatment (oral, inhaled or intranasal), current vitamin D supplementation other than that found in a daily multivitamin.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in FIT clinic at Columbia University Medical Center
* Ages 5-11
* obesity

Exclusion Criteria:Underlying disorder of bone metabolism

* chronic renal failure
* chronic steroid treatment
* current vitamin D supplementation other than that found in a daily multivitamin

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D level | 3 months after initiation of intervention
  A 25-hydroxyvitamin D level will be measured after 3 months of the intervention from a blood sample

SECONDARY OUTCOMES:
Waist circumference | 3 months after initiation of intervention
  Waist circumference will be measured after 3 months
Percentage body fat | 3 months after initiation of intervention
  Percentage body fat will be measured by bioelectrical impedance analysis 3 months after the intervention
Bone markers | 3 months after initiation of intervention
  Bone markers will be checked including PTH, osteocalcin, c-telopeptides, P1NP, alkaline phosphatase from a blood sample
Inflammatory markers | 3 months after initiation of intervention
  Inflammatory markers IL-6 and TNF-alpha will be checked from a blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Aviva B Sopher, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No